CLINICAL TRIAL: NCT02622009
Title: Human Rhinovirus and Respiratory Syncytial Virus From Bronchoalveolar Lavage and Bronchial Biopsies of Selected Patients With Stable Chronic Obstructive Pulmonary Disease.
Brief Title: Viral Infections in BAL and Bronchial Biopsies of Stable COPD Patients
Status: Completed | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Styliani Giannakaki, Resident in Respiratory Medicine, University of Athens
Other Study IDs: 10451
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: HRV and RSV Presence in the Lungs of Stable COPD Patients.
Keywords: stable COPD; bronchoalveolar lavage; biopsy; HRV; RSV
MeSH Terms: interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — BAL and bronchial biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- COPD I: BRONCHOSCOPIC PROCEDURE IN COPD PATIENTS STAGE I
  Interventions: Procedure: BRONCHOSCOPIC PROCEDURE
- COPD II: BRONCHOSCOPIC PROCEDURE IN COPD PATIENTS STAGE II
  Interventions: Procedure: BRONCHOSCOPIC PROCEDURE
- COPD III: BRONCHOSCOPIC PROCEDURE IN COPD PATIENTS STAGE III
  Interventions: Procedure: BRONCHOSCOPIC PROCEDURE
- NONSMOKERS: BRONCHOSCOPIC PROCEDURE IN NONSMOKERS
  Interventions: Procedure: BRONCHOSCOPIC PROCEDURE
- CURRENT OR EXSMOKERS: BRONCHOSCOPIC PROCEDURE IN CURRENT OR EXSMOKERS
  Interventions: Procedure: BRONCHOSCOPIC PROCEDURE

INTERVENTIONS:
Procedure: BRONCHOSCOPIC PROCEDURE — After the routine bronchoscopic inspection of the tracheobronchial tree, the investigators performed BAL from subsegmental bronchi and bronchial biopsies (3-4 per patient) from non infiltrated carina

SUMMARY:
Background: The presence of low-grade viral infection in the airways of patients with stable chronic obstructive pulmonary disease (COPD) could potentially have implications in the pathogenesis and progression of the disease, but previous studies have reported very different rates of human rhinovirus (HRV) and respiratory syncytial virus (RSV) genome detection in nasal and sputum samples. However, no study has investigated the presence of these viruses directly in the lungs by bronchoalveolar lavage (BAL) and bronchial biopsies. This study aimed to investigate whether HRV and RSV are present in the lungs of stable COPD patients by performing BAL and bronchial biopsies, and relate their presence with disease severity.

Methods: Consecutive patients with stable COPD and control subjects, who underwent diagnostic (e.g., lung cancer) and/or therapeutic (e.g., hemoptysis) fibreoptic bronchoscopy in a university hospital in Athens, Greece, were enrolled. The collected BAL and bronchial biopsies during bronchoscopy were subsequently processed for HRV and RSV RNA detection with real-time polymerase chain reaction (PCR). More specifically, the nucleocapsid gene and 5΄ non-coding region were searched for RSV and HRV detection, respectively.

DETAILED DESCRIPTION:
Patients and control subjects The population of the study consisted of consecutive patients with stable COPD and control subjects, who were referred to the investigators between October 2012 and November 2014 in order to undergo fibreoptic bronchoscopy for diagnostic (e.g., lung cancer) or therapeutic (e.g., hemoptysis) purposes. At study time, the clinical and functional status of COPD patients had been stable for at least 4 weeks, and none had received antibiotic treatment during the last 4 weeks. Exclusion criteria included atopic history, asthma, extensive pleural effusions, bronchiectasis, immunosuppression due to chemotherapy or systemic corticosteroids and all the contraindications of the bronchoscopic procedures. COPD severity was classified using postbronchodilator spirometric values according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines. Also, the patients were evaluated according to the combined COPD assessment. In this classification the impact of the disease on an individual patient is determined from the combination of the symptomatic assessment (CAT or mMRC scores), the patient's spirometric classification and/or the risk of exacerbations (number of exacerbations and history of hospitalization due to exacerbation in the preceding year).The control group was consisted of non-smokers or current/ex-smokers without COPD. The ex-smoking condition was defined as the cessation of smoking habit at least 1 year previously.

All the participants completed a questionnaire which included demographic characteristics and cigarette smoking status (pack/year). Τhe clinical status was evaluated according to the modified Medical Research Council (mMRC) scale of breathlessness and the Body mass , airflow Obstruction, Dyspnea, Exercise (BODE) index. Pulmonary function testing was performed and arterial blood gases and blood oxygen saturation by pulse oximetry in the sitting position were measured. Patients were asked about the number and the characteristics of the preceding exacerbations, the number and duration of preceding hospitalizations for respiratory disorders, their past medical history (asthma, allergy, sinusitis or nasal polyps), the presence of comorbidities (heart disease, malignancies, e.t.c.), and all the medication they used.

Both the COPD patients and control subjects were appropriately prepared (local anesthesia and intravenous sedation) in order to undergo transnasal fibreoptic bronchoscopy. After the routine bronchoscopic inspection of the tracheobronchial tree, the investigators performed BAL from subsegmental bronchi and bronchial biopsies (3-4 per patient) from non infiltrated carina.

All the samples were aliquoted, frozen and stored within 1 hour after sampling. HRV and RSV detection RNA samples were extracted from BAL and lung biopsies using the Maxwell 16 viral total nucleic acid (Promega). A Nucleocapsid (N) gene partial sequence, as well as a 5΄ non-coding region (5΄NCR) partial sequence were amplified for RSV and HRV, respectively.

Real-time PCR studies were performed. The primers/probes mix, that were used, have broad homology with a large range of HRV serotypes. Also, the primers/probes for RSV are able to distinguish RSV subtypes A and B whilst excluding the closely related human Metapneumoviruses. The primer and probe mix provided exploited the so-called TaqMan principle. A fluorogenic probe was included in the same reaction mixture which consisted of a DNA probe labeled with a 5'-dye and a 3'-quencher. Besides this, the probe was cleaved and the reporter dye and quencher were separated. The resulting increase in fluorescence could be detected on a range of real-time PCR platforms. Each time the kits were used, a positive and a negative control reaction were included in the run.

ELIGIBILITY:
Inclusion Criteria:

* stable COPD,indication for bronchoscopic procedure

Exclusion Criteria:

* atopic history, asthma, extensive pleural effusions, bronchiectasis, immunosuppression due to chemotherapy or systemic corticosteroids and all the contraindications of the bronchoscopic procedures

Ages: 51 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We enrolled 31 patients with COPD and 22 control subjects. The most common symptoms were dyspnea (32%), cough (19%) and hemoptysis (13%). Whereas 47% of participants did not mention any symptom, but referred to our department in order to investigate bronchoscopically abnormal radiographic findings revealed in chest computed tomography. The commonest comorbidities of COPD patients were arterial hypertension (47%), hyperlipidemia (20.7%) and coronary artery disease (17%), and of control subjects arterial hypertension (50%), hyperlipidemia (22,7%) and diabetes mellitus type 2 (13,6%).
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2010-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
HRV AND RSV PRESENCE | 7 days
  A Nucleocapsid (N) gene partial sequence, as well as a 5΄ non-coding region (5΄NCR) partial sequence were amplified for RSV and HRV, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: GEORGIOS ARSENIS, PROFESSOR, Study Director — University of Athens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Falsey AR, Formica MA, Hennessey PA, Criddle MM, Sullender WM, Walsh EE. Detection of respiratory syncytial virus in adults with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2006 Mar 15;173(6):639-43. doi: 10.1164/rccm.200510-1681OC. Epub 2005 Dec 30. PMID 16387798
- [Background] Seemungal T, Harper-Owen R, Bhowmik A, Moric I, Sanderson G, Message S, Maccallum P, Meade TW, Jeffries DJ, Johnston SL, Wedzicha JA. Respiratory viruses, symptoms, and inflammatory markers in acute exacerbations and stable chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2001 Nov 1;164(9):1618-23. doi: 10.1164/ajrccm.164.9.2105011. PMID 11719299
- [Background] Sethi S, Maloney J, Grove L, Wrona C, Berenson CS. Airway inflammation and bronchial bacterial colonization in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2006 May 1;173(9):991-8. doi: 10.1164/rccm.200509-1525OC. Epub 2006 Feb 10. PMID 16474030